CLINICAL TRIAL: NCT02472223
Title: Reducing Adenoviral Patient Infected Days
Acronym: RAPID
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: University of Alabama at Birmingham (Other); Illinois College of Optometry (Other); University of Illinois at Chicago (Other); Northeastern State University (Other); Ohio State University (Other); Massachusetts Eye and Ear Infirmary (Other); Brooke Army Medical Center (U.S. Federal Agency); University of California, Berkeley (Other); New England College of Optometry (Other); Massachusetts College of Pharmacy and Health Science (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 201412069
Record Dates: First submitted 2015-06-08; First posted 2015-06-15 (Estimated); Results first posted 2021-01-06 (Actual); Last update posted 2021-01-06 (Actual); Status verified 2021-01

CONDITIONS: Conjunctivitis; Adenoviral Conjunctivitis
Keywords: "Pink Eye"
MeSH Terms: conditions — Conjunctivitis | interventions — Povidone-Iodine; Lubricant Eye Drops; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Betadine 5% (Active Comparator): One time in-office administration (4-5 drops) of Betadine 5% limited to 2 minutes, followed by saline lavage.
  Interventions: Drug: Betadine 5%
- Artificial Tears (Placebo Comparator): One time in-office administration (4-5 drops) of artificial tears limited to 2 minutes, followed by saline lavage.
  Interventions: Drug: Artificial Tears

INTERVENTIONS:
Drug: Betadine 5% — One time in-office administration (4-5 drops) of Betadine 5% limited to 2 minutes, followed by saline lavage.
  Betadine 5% exposure to the ocular surface is limited to 2 minutes in-office administration, followed by saline lavage per labeling instructions.
  Other Names: Povidone Iodine
  Arms: Betadine 5%
Drug: Artificial Tears — One time in-office administration (4-5 drops) of artificial tears limited to 2 minutes, followed by saline lavage.
  Other Names: Saline Solution
  Arms: Artificial Tears

SUMMARY:
The primary aim of this pilot study is to generate data needed to design a definitive trial to compare the safety and efficacy of standard care with artificial tears vs. Betadine 5% (5% povidone-iodine) for the treatment of pink eye due to adenovirus. There is currently no FDA approved treatment for pink eye, a common and highly contagious eye infection caused by adenovirus. Standard care as recommended by the American Academy of Ophthalmology and American Optometric Association is instillation of artificial tears to relieve symptoms and possibly reduce the virus population. Betadine 5% is a commercially available, broad-spectrum antiseptic ophthalmic solution used for over 50 years to prepare the patient's eye and surrounding area for eye surgery. Because Betadine 5% kills bacteria and viruses, it may be useful in treating adenoviral conjunctivitis. Betadine 5% is inexpensive, safe, widely available, and immune to the development of bacterial/viral resistance. Betadine 5% has the potential to significantly impact the clinical management of "pink eye" worldwide.

This pilot study has received funding from the National Eye Institute. Participants who meet eligibility criteria will be randomized using a masked randomization packet to receive one-time, in-office treatment with either artificial tears or Betadine 5%.

Patients who agree to study participation will answer questions about their pink eye symptoms, medical and ocular history, have an eye examination and be tested to confirm "pink eye" due to adenovirus using a FDA approved "point of care" immunoassay. Participants testing positive for adenovirus will have a tear sample taken to measure viral load by qPCR. Randomization and a one-time treatment with either (standard care) artificial tears or Betadine 5% will be done on the first visit. Follow-up visits are at 1,4,7,14 and 21 days. At each visit, symptoms of pink eye are asked, a standardized study eye examination is given by the masked clinician and a sample of tears is taken to assess viral load by qPCR.

DETAILED DESCRIPTION:
Aim 1: To compare the safety and efficacy of 5% Betadine to artificial tears in reducing viral load in patients with adenoviral conjunctivitis.

Aim 2: To compare the efficacy of 5% Betadine to artificial tears in reducing patient reported bothersomeness of ocular symptoms.

"Pink eye" (adenovirus conjunctivitis Ad-Cs)is a common ocular condition, with afflicted patients comprising as much as 2% of a general practitioner's practice. Partly due to the ability of adenovirus to remain infectious in the desiccated state for weeks at room temperature, Ad-Cs is more contagious than other forms of conjunctivitis and it can be spread via both ocular or respiratory secretions. Owing to the highly contagious nature of this condition, Ad-Cs outbreaks occur where people congregate: schools, military units, nursing homes, workplaces, community and health-care facilities. With respect to the latter, the nosocomial spread of the condition is a significant public health issue as 17% of 145 cases, 44% of 192 cases and 85% of 132 cases were reported to originate at the place of eye examination. The infection spreads from the first affected eye to the fellow eye in a majority of patients, and secondary transmission of viral conjunctivitis to members of the same household is estimated to occur at a rate of 20%. Outbreaks of Ad-Cs spare no nationality, age, gender or social class and because of the epidemic potential of some adenoviral serotypes, Ad-Cs is a reportable condition in Germany and Japan. A treatment that decreases the duration of the infectious period could have substantial impact in reducing the spread of Ad-Cs outbreaks.

To insure timely completion of recruitment, especially since outbreaks are seasonal and episodic, the study has recruited 6 participating clinical sites nationally. To attain the overall sample target of 50 randomized patients, about 200 pts with pink eye will need to be screened. Each clinic will screen 30-40 patients and randomize 8-10 over a 12 month period.

Patients who present with presumed acute Ad-Cs, who are 19 years of age or older and report symptom onset of 4 days or less in the first affected eye will be invited to undergo eligibility screening.

Over a 12 month recruitment period, 10 Clinical Centers will screen at least 200 patients who present with presumed Ad-Cs, to enroll a target sample of 50 eligible patients. 10 Clinics include Illinois College of Optometry, Ohio State University, Northeastern State University and University of Alabama at Birmingham, Brooke Army Medical Center, University of California, Berkeley, Massachusetts Eye and Ear, New England College of Optometry, University of Illinois and Washington University School of Medicine. These clinics provide geographic diversity and multi-ethnic representation (including African American, Asian, Caucasian, Hispanic and Native American groups). Because patients with pink eye are more likely to see an optometrist than an ophthalmologist, PI's of Clinics are optometrists.

Patients who consent to participation:

* Participant completes eligibility screening about 30 minutes - confirmation of age and symptom duration, a symptom survey, an eye examination;
* AdenoPlus(TM) test to confirm adenoviral conjunctivitis (Screening/Baseline Form);
* Participants who test positive by AdenoPlus(TM) are "fully eligible" and a tear sample will be taken for qPCR testing.

Fully eligible participants

* Will be randomized using masked packets identified by serial numbers containing the randomized treatment with either artificial tears or Betadine 5%;
* "Treating" unmasked study certified clinician will administer treatment as randomized;
* Participants will rate the discomfort of treatment to assess treatment tolerability and asked to guess whether they received artificial tears or Betadine 5%.

Follow-up visits will be scheduled for 1, 4, 7, 14 and 21 days after randomization. Each follow-up visit is about 30 minutes.

* Participants will rate the discomfort of treatment to assess treatment tolerability on day 1 post treatment;
* Masked clinician/technician will ask the 10-question pink eye ocular symptom questionnaire;
* Masked clinician will perform the eye examination;
* Masked clinician/technician will take conjunctival tear sample for analysis of viral load by qPCR.
* Participants who miss f/up visits will be asked to complete the symptom checklist by telephone or by secure REDCap data entry.

All study-related encounters with potential study participants will be conducted in private, closed-door, "Red Eye" examination room in the clinical center. All study certified personnel will ensure patient confidentiality at all times. The minimum amount of information needed for the study will be collected from study participants. All research study data are coded as to clinic site and patient ID and do not include personal health data. Personal health data are kept physically separate from research study data. All data are kept in HIPAA compliant office spaces. All study data will be collected and maintained using a secure, password protected web-based data capture program (REDCap).

The study drug, Betadine 5% is FDA approved for topical ocular surface application to the cornea, conjunctiva and palpebral fornices and is used in this study at the recommended dose, age group, duration and method of application. Risk is minimized by limiting administration to a single, one-time, in-office application. A study certified optometrist/technician instills artificial tears or Betadine 5% in the study eye. If there are immediate untoward reactions, the patient is in a fully equipped and staffed eye care facility where appropriate expertise and treatment are available. Participants are closely monitored with follow-up eye examinations at 1, 4, 7, 14 and 21 days after treatment.

Potential nosocomial infections are minimized by asking the patient to use hand sanitizer before entering the examination room. Patient signs only the consent form and all other surveys are administered by the clinician/technician. We will observe strict adherence to current CDC disinfection protocol for Ad-Cs. Patients reporting marked symptoms will be withdrawn from the study and managed according to standard clinical care guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Age: Patients will be 18 years and older.
* Duration of pink eye symptoms: No more than 4 days in first affected eye Positive immunoassay test "AdenoPlus(TM)" for presence of adenovirus.
* Sex: "Pink eye" {adenoviral conjunctivitis (Ad-Cs)} occurs with equal prevalence in males and females, therefore we will recruit both genders.
* Race/Ethnicity: Individuals of all races and ethnicities will be invited to participate in this study. Patient recruitment will reflect the distribution of race/ethnicity demographics for the patient population specific to each study site.

Exclusion Criteria:

* Patients with history of herpes simplex infection or corneal ulceration
* Eye surgery in the last 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2015-03-23 (Actual); Primary Completion 2018-06-01 (Actual); Study Completion 2018-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mae O Gordon, PhD, Study Chair — Washington University School of Medicine
Locations (1):
- Mary Migneco, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified patient data will be shared. Request for data access should be sent to Mae Gordon mae@wustl.edu.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: July 2023
Access Criteria: Data Access Request will be reviewed by the Steering Committee.

REFERENCES:
- [Derived] Morettin CE, Harthan JS, Huecker JB, Perera CD, Than T, Whiteside M, Johnson SD, Shorter E, Migneco MK, Olson CK, Alferez CS, Camp D, Hartwick ATE, Gordon MO. Correlation of Adenoviral Titers with Severity of Adenoviral Conjunctivitis and Time to Viral Clearance for 21 Days. Optom Vis Sci. 2023 Mar 1;100(3):187-193. doi: 10.1097/OPX.0000000000001999. Epub 2023 Feb 7. PMID 36749104
- [Derived] Whiteside MM, Shorter ES, Margolis MS, Alvi F, Huecker JB, Than TP, Migneco MK, Harthan JS, Morettin CE, Hartwick ATE, Johnson SD, Perera CD, Gordon MO. Success of Masking 5% Povidone-Iodine Treatment: The Reducing Adenoviral Patient Infected Days Study. Optom Vis Sci. 2021 May 1;98(5):469-475. doi: 10.1097/OPX.0000000000001691. PMID 33973917

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants, who are ≥ 18 years of age and report symptom in the first affected eye onset ≤ 4 days, will be informed of the study by Clinical Center personnel and asked if they would be interested in learning more.
Period: Overall Study
Arm/Group | Betadine 5% | Artificial Tears
Started | 16 | 12
Completed | 10 | 7
Not Completed | 6 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Betadine 5% | Artificial Tears | Total
Number analyzed (Participants) | 16 | 12 | 28
Age, Categorical [Count of Participants; unit: Participants] — Population: We only analyzed those participant who were qPCR positive.
  Participants
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 15 | 11 | 26
    >=65 years | 1 | 1 | 2
Sex: Female, Male [Count of Participants; unit: Participants] — Population: We only analyzed those participant who were qPCR positive.
  Participants
    Female | 8 | 7 | 15
    Male | 8 | 5 | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: We only analyzed those participant who were qPCR positive.
  Participants
    Hispanic or Latino | 3 | 2 | 5
    Not Hispanic or Latino | 13 | 9 | 22
    Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: We only analyzed those participant who were qPCR positive.
  Participants
    American Indian or Alaska Native | 4 | 1 | 5
    Asian | 1 | 0 | 1
    Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
    Black or African American | 7 | 4 | 11
    White | 3 | 5 | 8
    More than one race | 0 | 1 | 1
    Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants] — Population: We only analyzed those participant who were qPCR positive.
  Participants
    United States | 16 | 12 | 28

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Peak Viral Load
Description: To compare efficacy of Betadine 5% to artificial tears to change from peak viral load in Adenoviral conjunctivitis
Time Frame: 21 days
Population: Subgroup of 16 patients randomized to Betadine and 12 patients randomized to artificial tears who tested positive for adenoviral conjunctivitis by qPCR at baseline. Viral load was assessed at baseline, post treatment follow-up days at 1-2, 4-5, 7, 14 and 21.
Measure: Median (Full Range); unit: Percent of peak Viral Load
Arm/Group | Betadine 5% | Artificial Tears
Number analyzed (Participants) | 16 | 12
Percent of peak Viral Load | 1.9 [0 to 7.6] | 13.2 [1 to 32.3]
Statistical Analysis 1: Comparison: Betadine 5% vs Artificial Tears; Test type: Superiority; p = 0.02, Wilcoxon (Mann-Whitney) — p-value is not adjusted for multiple comparisons; Median Difference (Final Values) = 90

2. Secondary Outcome: Participant Reported Bothersomeness of Ocular Symptoms
Description: Participants reported bothersomeness of ocular symptoms on a 10 point scale 0=not at all. 10=very bothersome
Time Frame: 21 days
Population: Patient reported bothersomeness of ocular symptoms was assessed at baseline, post treatment follow-up days at 1-2, 4-5, 7, 14 and 21.
Measure: Median (Full Range); unit: Unit on a scale
Arm/Group | Betadine 5% | Artificial Tears
Number analyzed (Participants) | 16 | 12
Unit on a scale | 4.5 [0 to 10] | 8.0 [0 to 10]

ADVERSE EVENTS:
Time Frame: Adverse event data was collected during the full length of follow-up, which was 21 days.
Groups:
- Betadine 5%: One time in-office use (4-5 drops)
  Betadine 5%: One-time, in-office administration of Betadine 5%.
  Betadine 5% exposure to the ocular surface is limited to 2 minutes in-office administration, followed by saline lavage per labeling instructions.
- Artificial Tears: Standard of Care
  Artificial Tears: Standard of care
Arm/Group | Betadine 5% | Artificial Tears
All-Cause Mortality (participants affected / at risk) | 1/16 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/12
Other Adverse Events (participants affected / at risk) | 0/16 | 0/12

LIMITATIONS AND CAVEATS:
Small pilot study. Sample consisting of only adults. Lost to follow-up. High false positive rate of point-of-care immunoassay which necessitated a modified intention-to-treat analysis of participants with PCR confirmed Ad-Cs.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2020-04-23): https://cdn.clinicaltrials.gov/large-docs/23/NCT02472223/Prot_SAP_ICF_000.pdf